CLINICAL TRIAL: NCT05977491
Title: Randomized Controlled Trial in Nepal: Introducing Point-of-care Tests and Identifying Barriers to Reduce Antibiotics for Vaginal Discharge
Brief Title: Point-of-care Tests for Vaginal Discharge in Nepal
Acronym: POCT-BRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Kathmandu University School of Medical Sciences (Other); University of Oslo (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 335889
Record Dates: First submitted 2023-07-04; First posted 2023-08-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Vaginal Discharge; Sexually Transmitted Diseases
Keywords: antibiotic overtreatment; psychosomatic; domestic violence; anxiety and depression; chlamydia trachomatis; neisseria gonorrhoea; trichomonas vaginalis; bacterial vaginosis; process evaluation; point-of-care-test
MeSH Terms: conditions — Vaginal Discharge; Sexually Transmitted Diseases; Anxiety Disorders; Depression; Vaginosis, Bacterial | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Three armed RCT.
  1. Standard treatment
  2. POCT result based treatment
  3. POCT result based treatment plus patient education and addressing of anxiety, depression and domestic violence
Who Masked: Participant, Outcomes Assessor
Masking Description: The health care provider will know if informed about the POCT results (in groups 2,3) or not (group 1). He will not know if patient is in group 2 or 3.
  The investigator will be present at various times during inclusion for quality control and therefore is not blinded.
  The outcome assessor ( the PhD candidate and the statistician) will receive data files without specific group label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard treatment (No Intervention): Patients are treated by the health care practitioner according to local protocol. This protocol corresponds to the syndromic approach without laboratory or microscopic testing. This may or may not include inspection and examination of the vulva, vagina, cervix and lower abdomen.
- POCT based treatment (Active Comparator): The health care practitioner is informed about the POCT results for CT and NG (positive or negative). In addition, if the pH is within the normal level (4.5 and below). If it is higher, he will receive the outcome of the whiff test (positive or negative). For the second half of enrolled participants: if pH is > 4.5 and whiff test is negative, the OSOM test for TV will be performed an self collected vaginal discharge. The Health care practitioner is informed if the TV test is positive or negative.
  Examination of the patient is performed according to the discretion of the health care practitioner.
  Interventions: Diagnostic Test: Health care practitioner is informed of POCT results for CT and NG; Diagnostic Test: Health care practitioner is informed about POCT result for TV and BV
- POCT based treatment PLUS (Active Comparator): Same as in POCT based treatment PLUS in addition:
  1. All women complete a questionnaire prior to examination, including a screening tool for anxiety and depression and domestic violence. If they screen positive, they are offered psychological counseling. All women are informed about referral possibilities to a crisis management center.
  2. Patients are given a short educational leaflet and 10 min audio-recording about physiological and abnormal vaginal discharge and about problems associated with unnecessary use of antibiotics.
  Interventions: Diagnostic Test: Health care practitioner is informed of POCT results for CT and NG; Diagnostic Test: Health care practitioner is informed about POCT result for TV and BV; Other: addressing psycholsocial problems

INTERVENTIONS:
Diagnostic Test: Health care practitioner is informed of POCT results for CT and NG — Molecular, PCR based near-POCT performed by the research assistant on self -collected urine. The outcome is positive or negative
  Other Names: GeneXpert test from Cepheid for CT andNG
  Arms: POCT based treatment; POCT based treatment PLUS
Diagnostic Test: Health care practitioner is informed about POCT result for TV and BV — The pH of vaginal secretion is measured from a self-collected swab by the research assistant, and if above 4.5 a dropp of KOH is added. If it smells fishy, the whiff test is positive.
  Other Names: Narrow range pH and confirmatory whiff test with potassium hydroxide (KHO), Amsel criteria; for second half of participants to be included: if pH > 4.5 and whiff test is negative, the OSOM test will be performed for TV
  Arms: POCT based treatment; POCT based treatment PLUS
Other: addressing psycholsocial problems — 1. Participants screening positive for anxiety, depression or domestic violence will be offered psychological counseling or referral to a crisis management center in the POCT-PLUS arm
  2. All participants of the POCT-PLUS arm receive audio- visual and written education on vaginal discharge and antibiotics
  Other Names: providing basic information on vaginal discharge and antibiotics
  Arms: POCT based treatment PLUS

SUMMARY:
The goal of this clinical trial is to examine if and how the implementation of point-of care-tests (POCT) for sexually transmitted infections in the management of abnormal vaginal discharge reduces the overtreatment with antibiotics in a low income country. The setting is a university hospital in a semi-rural area in Nepal and several of its rural out-reach-centers. The plan is to include 1500 women attending the gynecological outpatients with a problem of vaginal discharge over approximately a one year period.

The main questions the clinical trial aims to answer are:

* Does POCT guided treatment result in reduced over-treatment of antibiotics, compared to the current approach in Nepal?
* What are the barriers and facilitators of the acceptability of POCTs and the resulting treatment from the perspective of both patients and health care practitioners?

Participants will be randomized in three groups:

* standard treatment according to current practice
* POCT result based treatment
* POCT result based treatment plus patient education and addressing of psycho social vulnerabilities

DETAILED DESCRIPTION:
Abnormal vaginal discharge (AVD) is a common problem women seek treatment for allover the world. In low and low- middle income countries (LLMICs) about one third of these women will have a sexually transmitted disease (STI) caused by Chlamydia trachomatis (CT), Neisseria gonorrhoea (NG) or Trichomonal vaginalis (TV). Approximately another third will have an imbalance in the vaginal microbiotic flora, bacterial vaginosis (BV). These women and their sexual partners in the case of sexually transmitted diseases will benefit from specific antibiotic treatment. The last third of women will not have any infection and there are indications that psychosocial problems may be expressed as somatic complaints, for example of abnormal vaginal discharge in some cultures.

In high income countries, with the help of laboratory-based tests, available after few days, treatment is usually with a narrow spectrum antibiotic for specific bacteria. This involves less risk for the development of antibiotic resistance. In low-income countries, laboratory testing is not feasible due to costs and logistics. Women are usually receiving antibiotic treatment with several types of antibiotics to cover STIs. More recently, point-of -care tests which are nearly as accurate as laboratory-based tests have been developed. Implementation studies for these tests in LLMICs are lacking. However, these molecular tests are still expensive.

In this study the investigators propose a combination of molecular tests for the two most serious infections (CT and NG) and a cheap and simple tests for TV and BV, which both are treated with the same type of antibiotic.

In addition, women attending an outpatient department in a LLMIC setting, expect (antibiotic) treatment, which they will not receive with a negative POCT. In LLMICs it is common practice to purchase over the counter medication, inclusive antibiotics. In particular for women with negative POCT results, there could be a lack of adherence to treatment recommendations.

We want to examine the following research questions (RQ) in the context of treatment for vaginal discharge:

1. Can POCTs effectively reduce the use of antibiotics? A) The amount of antibiotics prescribed at the time of the appointment B) the proportion of correcly pescribed antibiotics (as defined by gold-standard tests) C) Additional antibiotics used, as reported by the patients,
2. Barriers and facilitators for patients and health practitioners with a focus on psychosocial and educational elements

For this purpose, a RCT with three arms was designed:

(A) Treatment as usual, (B) Treatment according to POCT results, (C) Treatment according to POCT results and additional patient information on vaginal discharge and antibiotics and screening and available counseling for psychosocial problems.

The investigators plan to include 1500 women with the complaint of abnormal vaginal during a 10-12 month period at Dhulikhel hospital, a tertiary university hospital in central Nepal and selected outreach centers in 2024 and 2025.

Sample size calculation are based on RQ1 and RQ2, feasibility of recruitment and the precision of the estimates, a two-sided 95 % confidence intervals (CI). For RQ1, the use of any antibiotics will be assessed in both POCT arms combined versus the treatment as usual arm (n = 1500), whilst the effect of the educational material on the use of over-the-counter medications will be assessed in the POCTplus versus the POCT group (n = 1000). As many as 85% of women with AVD are over-treated with antibiotics in LLMICs, around 50 % receive antimicrobial resistance driving antibiotics and it is expected, that around 40 % women in the POCT group will subsequently seek over the counter antibiotics. With 1500 participants randomized 1:1:1, a 10 to 20 percentage point reduction in any of these measures will produce CIs with a width between 8 and 12 % and at least 90% power. When allowing for around 40 % loss to follow-up, when assessing the use of over-the-counter antibiotics, the expected width of the CI is still around 15 %.

The investigators will collect self-sampled urine and vaginal swabs from all included women and a self-administered questionnaire with a color-coded audio-computer. The questionnaire contains demographic information and a validated tool to screen for anxiety, depression and domestic violence.

Gold standard testing for the STIs and BV will be performed on all women. Participants will be randomized into three arms. In the standard treatment arm, the attending health practitioner will not be informed about POCT results. In the two POCT arms, the health care practitioner will be informed about CT and NG status and about the pH, inclusive a confirmatory whiff test.

Addition (22.09.2024): after the first 100 participants it was recognized, that sensitivity of the combination pH and whiff test was unacceptably low for TV for women with a high pH and negative whiff test. We will add another low cost, immunological POCT for TV for women with a high pH and a negative whiff test after the first half of participants has been enrolled. Based on our additional power calculation, we will have sufficient power to seperately analyse the diagnostic accuracy for TV both before and after the addition of this test.

In the POCT-PLUS arm, patients will receive additional educational information about physiological and abnormal vaginal discharge and about potentially negative effects of antibiotic treatment. In this arm, woman screening positive for positive for anxiety, depression or domestic violence will be offered psychological counseling or referral to a crisis center Participants will be followed up telephonically after 1 and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting with vaginal discharge to gynecological outpatients

Exclusion Criteria:

* Minors below the age of 18 years.
* Any bleeding from the vagina.
* Suspicion of gynecological cancer.
* Previous inclusion in the same study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Vaginal discharge under investigation is restricted to genetic females.
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants overtreated with antibiotics (excluding antifungals) | At inclusion
  Comparing the proportion of women overtreated with antibiotics for treatment depending if the health care practitioner was informed about the POCT results (arm 2+3) or not (arm1). Reported by the health care practitioner. Overtreatment is defined as receiving a cephalosporin when NG is negative; a tetracycline when CT is negative; a macrolide when NT and CT are neagtive; a nitroimidazole when the gold standard test for TV or BV is negative.
  These subgroups are anlayzed: (a) before addition of an additional POCT for women with a pH above 4.5 and a negative whiff test, this is the first half of participants; (b) after addition of this extra test, for the second half of included participants; (c) suburban- and (d) rural clinics.
  We compare arm 1 with the combined arms 2+3.
Proportion of participant prescribed antimicrobial resistance driving antibiotics | At inclusion.
  Comparing the proportion of women in arm 1( comparison arm) compared to arm 2 and 3 (intervention arms), receiving AMR driving antibiotics (Cephalosporins, Azithromycin, Ciprofloxacillin), depending if the health practitioner received POCT results.
  These subgroup analysis are planned: (a) suburban vs urban clinics. We compare arm 1 with the combined arms 2+3.
Proportion of participants adhering to treatment recommendations | At telephonic follow up after 1 month.
  Among participants, where the health practitioner had received POCT results, we compare the proportion of women adhering to treatment recommendations, depending on if they received psycho social intervention (arm 3) or not (arm2), in the arm Adherence is defined as follows: (1) participants report they took the prescribed medication, (2) no additional purchase of antibiotics; (3) no purchase of other medication for VD.
  Subgroup analysis for (a) suburban and (b) rural areas. (c) participants screening positive for domestic violence or (d) anxiety or depression, offered counseling or not.
  We compare all arms (arm1, 2 and 3)

SECONDARY OUTCOMES:
Proportion of participants prescribed antibiotics | At inclusion
  Comparing the proportion of participants prescribed antibiotics depending if the healthpractitioner was informed about POCT results or not. Comparing arm 1 versus arm 2+3.
  Following subgroup analysis: (a) first half of participants before adding another POCT for TV; (b)second half of participants after adding TV POCT; (c) suburban-; (d) rural clinic.
  (e) 8 antibiotic groups: tetracyclines (including doxycillin), kinolones (ciprofloxacin), macrolides (erythromycin, azitromycin), sulfonamides (trimethoprim(-sulfa), imidazolderivates (metronidazole), penicillins(including Selexid), cephalosporines, other antibiotics.
Undertreatment with antibiotics for CT, NG, TV and BV with or without POCT guided treatment | At inclusion
  We compare proportions of participants under treated for CT, NG, TV or BV, depending on , if the health practitioner received POCT results or not.
  Definition: of under treatment: not receiving a tetracycline or macrolide with a positive CT test, no Cephalosporin with positive Ng test, no imidazoles with a positive gold standard test for TV or BV. We compare control groups (arm 1) with the intervention groups (arm 2+3)
Proportion of women adhering to treatment recommendationss | At telephonic follow up 4 months after initial consultation
  Description: Among participants, where the health practitioner had received POCT results, we compare the proportion of women adhering to treatment recommendations, depending on if they received psycho social intervention (arm 3) or not (arm2), in the arm Adherence is defined as follows: (1) participants report they took the prescribed medication, (2) no additional purchase of antibiotics; (3) no purchase of other medication for VD. Subgroup analysis for (a) suburban and (b) rural areas, participants screening positive for (c) domestic violence, (d) anxiety or depression, offered counseling or not.
  We compare all arms (arm 1, 2 and 3).
Does educational and psychosocial measures affect change in VD symptoms? | At telephonic follow up after 4 weeks and 4 months.
  Comparing graded VD symptoms (3 grades), depending on if participants received educational material or psychosocial measures (in arm 3)? Subroups: (a) participants screening positive for domestic violence , (b) participants screening positive for anxiety and/or depression, (c) participants receiving counseling for anxiety and depression Overall comparison arm 1,2,3.
  -
Comparing prevalence of screening positive for anxiety and depression before and 4 months after consultation for VD | At telephonic follow up, 4 months after initial consultation
  Change in proportion of participants screening positive for anxiety or depression 4 months after consultation for VD
Comparing mean patient satisfaction with consultation and treatment between all RCT arms | At follow up after 4 months
  Satisfaction with (a)consultation and (b) treatment is measured on a self-reported scale from 1-5 at the telephonic follow up interview. We will compare mean (SD) for all three arms

OTHER OUTCOMES:
Prevalence STIs and associated demographic and clinical findings | at enrollment
  Relative risk of Chlamydia trachomatis, Neisseria gonorrhoe, Trichomonas vaginalis and bacterial vaginosis in relation to age (three age groups), socioeconomic status (4 categories), suburban- or urban population, reproductive history (parous, condom use, vaginal douching), subjective symptoms (pain or not) and clinical findings ( abnormal findings or not) All groups regardless RCT arm are included
Associations between self reported domestic violence, anxiety and depression and STI diagnosis | at enrollment
  Domestic violence is measured by the module of the Nepal Demographic Health survey 2016, which is the Nepalese adaptation of the Conflict Tactics Scale, binominal outcome.
  Anxiety and depression symptoms are measured with the Hopkins symptom check list, there is a cut off on an continuous scale, thus it can be used also as a binominal variable. We will perform cross tabulations with risk estimation for (a) STI diagnosis and a positive anxiety and depression score; (b) STI diagnosis and screening positive for domestic violence and (c) screening positive for anxiety and depression and domestic violence.
Diagnostic accuracy for bacterial vaginosis(BV) and/or Trichomonas Vaginalis (TV) with pH and whiff test | First 500 participants at Dhulikhel Hospital and first 250 participants at ORC.
  All groups, independent randomization. PH >4.5 and a positive whiff test from a self- collected vaginal swab is defined as positive for BV or TV. Compared to gold standard tests from selv- collected urine: Nugent scoring for BV and molecular test (GenExpert, Cepheid) for TV.
  Sensitivity, specificity, positive and negative predictive value are calculated.
Diagnostic accuracy of sequential screening for bacterial vaginosis (BV) and /or Trichomonas vaginalis (TV) | Second half of participants at Dhulikhel Hospital (participant 501 - 1000) and out-reach -centers (participantn1251-1500).
  All participants independent of RCT arm are included. If Ph is > 4.5 and whiff test of self-collected vaginal swab is positive, the participant is defined positive for BV or TV. If the ph is 4.5 or lower the participant is considered negative for BV and TV. If pH is >4.5 and whiff test negative, a lateral flow test (OSOM test) is performed on self-collected vaginal discharge. If this test is positive, the participant is considered TV positive and BV negative. if this test is negative, the participant is considered TV and BV negative. Compared to gold standard test for TV GenExpert (self-collected urin), and for BV Nugent scoring from self-collected vaginal discharge.
  We calculate sensitivity, specificity, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: Risa AM Lonnee-Hoffmann, PhD, Principal Investigator — Norwegian University for Science and Technology
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Kavre, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the applicable article, after deidentification (without participant number) (text, tables, figures,and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. For five years
Access Criteria: To researchers who submit a sound proposal. Proposals should be directed to risa.lonnee-hoffmann@ntnu.no. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Linkto be included).
URL: http://dataarkivering.sikt.no/

REFERENCES:
- [Derived] Shrestha S, Shakya S, Infanti JJ, Skovlund E, Simpson MR, Lonnee-Hoffmann RAM. Implementing point-of-care tests to optimize antibiotic use for vaginal discharge: a study protocol for a randomized controlled trial in Nepal. Trials. 2025 Dec 12. doi: 10.1186/s13063-025-09333-4. Online ahead of print. PMID 41388307